CLINICAL TRIAL: NCT05549648
Title: Artificial Intelligence-Based APP for Home Oral Muscles Exercises for Healthy Adults
Brief Title: The Oral Biomechanical Functions of Hong Kong Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UW21-324
Record Dates: First submitted 2022-07-13; First posted 2022-09-22 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2022-08

CONDITIONS: Oral Manifestations
Keywords: oral frailty; oral muscle; home oral exercise
MeSH Terms: conditions — Oral Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-controlled Study (Other): Hong Kong citizens over 50 years old
  Interventions: Other: Home oral excrise

INTERVENTIONS:
Other: Home oral excrise — The current study aimed to evaluate the efficacy and user experience of mobile phone APP, a mobile application with AI component in facial movement tracking, in improving oral functions of elderly people

SUMMARY:
Hong Kong and Japan are similar in terms of facing the super-ageing society. Maintaining oral function in elderly is particularly important because it affects social, physical and mental health to the people and to the society. By using technology seems to be one of the solutions in dealing with this. Thus, this project aims at using state-of-the-art Age-tech that have been used in Japan to implement "Oral Frailty" concept in Hong Kong. Through identifying oral biomechanical in elderly population, the investigators expect the situation can be improved, and the data analysed and collected can be useful and impactful that can influence the dental communities around Southeast Asia and the globe.

DETAILED DESCRIPTION:
In 2020, this is not only a year of pandemic but also the year that the number of "super-aged" countries - where more than one in five of the population is 65 or older - reach to 13 including Japan, Germany, Italy, Netherlands, France, Sweden, Portugal, Slovenia and Croatia. By 2030, the number of countries would increase to 34 including Hong Kong, Korea, the US, the UK and New Zealand [1]. These countries are currently generating 80% of global GDP [2]. So, this 10-15% of super-aged global population is expected to create economic burden around 13-20% of GDP depending on the countries and policies [3], that will indeed severely affect global economy in the future if the ageing problem is not properly treated.

Hong Kong and Japan ranks number 1 and 2, respectively, lowest in 0-14 children population in the high income countries/region [2]. Facing to this low birth rate, according to the "Hong Kong Population Forecast 2020-2069", by 2069, the number of elderly people aged 65 or over in Hong Kong will reach 2.6 million, accounting for about 35.9% of the total population. The labor force between the ages of 15 and 64 will shrink to 3.9 million, accounting for 54.6% of the population [4].

In particular to dentistry, maintaining the oral function in elderly is very important, due to:

1. food nutrients - when you eat you can obtain the nutrients from food, this provides you the essential energy for daily life. Loss of teeth or misfit of artificial teeth positively correlated with the risk of development in general chronic diseases [5].
2. self-esteem - oral appearance and communication are significant factors contributing to elderly's psychological well-being and social life, impacting to the oral health related quality of life (OHRQoL) [6].
3. neurological disorder - oral health was shown to related with strokes [7] and Alzheimer's disease [8] due to the invasion of oral bacteria such as Aggregatibacter actinomycetemcomitans, Prevotella intermedia, and Porphyromonas gingivalis. Only these two neurological disorders have accounted 0.08-0.52% loss of GDP in 47 prefectures in Japan in 2012, and the GDP lost is forecasted to be increasing continuously [9]. Tooth lost is a key factor.

Apparently, oral health is important to have healthy aging. The dental personnel play a key role in oral health, in terms of prevention, intervention, and education. In particular, prevention and education are comparatively low-cost strategies while intervention bears the higher cost, as shown in our previous study that countries/regions with better economic status had fewer severe impacts on diet-related aspects of OHRQoL [10]. Besides, our study also showed social and physiological factors "trouble pronouncing words" ranks significantly high similarly as other dietary factors, i.e., "uncomfortable to eat", "diet unsatisfactory" and "interrupt meals" among the developed countries with high economy. Indeed, the loss of teeth, new dental prostheses, and oral muscle dysfunction due to aging are the major contributing factors of pronunciation trouble. This physiological "oral frailty" declines the elder's mental and social health, and should be identified and addressed before the need for long-term care [11].

Utilizing technology to understand this situation deemed possible and "Age-tech" becomes an essential part of health technologies which means applying technology to identify, improve and treat oral frailty situations. The technology can also be useful to monitor and evaluate the efficiency of oral health conditions during this pandemic when the patients have limited mobility around the society.

ELIGIBILITY:
Inclusion Criteria:

* Population with aged (50-90 y.o.) neurologically healthy citizens in Hong Kong who have at least 1 occluding paired molars.
* Can read Traditional Chinese and communicate in Cantonese
* Possessed a smartphone with internet access and was able to use it on their own or with the help of at least one family member
* passed the Montreal Cognitive Assessment 5-Minute Protocol (Hong Kong Version)

Exclusion Criteria:

* Subject who was under 50 or unable to give consent.
* Subject who has Cerebrovascular accident, Head and Neck Cancers, Neurologic Diseases, and other severe systemic diseases.
* Subject who is receiving radiotherapy and chemotherapy.
* Subject who was medically unfit.
* Subject who has no molar.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Occlusal force assessment | The 1, 30, 90, and 120 days after recruitment. The investigators wanted to see if exercise would help oral muscle performance, there's a lack of data on this, so the investigator couldn't determine a change over time.
  The tooth models and occlusion will be taken to record the occlusal contact point, area and distribution, by intra-oral scanner (CEREC Omniscan / 3Shape), which is a standard practice at HKU. The occlusal force (N), occlusal contact area (mm2), maximum occlusal pressure (MPa), average occlusal pressure (MPa) of both sides are measured respectively, using occlusal pressure measurement film (Dental Prescale® II 50H, GC Corp) that is scanned with a dedicated scanner (GT-X830, Epson) with analysis software (Bite force analyzer, GC Corp).
Masticatory efficiency | The 1, 30, 90, and 120 days after recruitment. The investigators wanted to see if exercise would help oral muscle performance, there's a lack of data on this, so the investigator couldn't determine a change over time.
  Gluco sensor (GS-II, GC Corp) will be used to quantitatively analyze the chewing ability
  1. Rinse mouth for 3 times, 20s at least for each time.
  2. Insert the test stick into GS-2, power on, and wait 6 seconds.
  3. Chewing for 20s, use the preferred chewing side.
  4. Rinse mouth with 10ml pure water and spit into the paper cup with a blue filter.
  5. Discard the jelly residue in the filter, mix up the liquid (10s), dip the solution with a micro brush, point it on the test stick, wait for 6s for result reading, record reading: the concentration of sugar: ____mg/dL.
Tongue function assessment | The 1, 30, 90, and 120 days after recruitment. The investigators wanted to see if exercise would help oral muscle performance, but there's a lack of data on improving this function, so the investigator couldn't determine a change over time.
  Tongue pressure sensor (TPM-02, GC Corp) which indicates the tongue physical function, will be used to record the maximum tongue pressure (MPa) for 3 times of each participant, then tongue endurance will also be measured for 3 times by determining how long tongue could sustain 60% of their maximal pressure.
Dry mouth | The 1, 30, 90, and 120 days after recruitment.
  A Chinese (Cantonese) version of dry mouth questionnaire consisting of 8-item xerostomia questions with a maximum total score of 32 points was used for subjective assessment, using a Likert format rated on a 4-point scale (1 not at all, 4 very much). Participants graded each aspect, with a higher score indicating impaired salivary function
Oral health-related quality of life | The 1, 30, 90, and 120 days after recruitment.
  The Chinese-validated version of the Oral Health Impact Profile-14 (OHIP-14) questionnaire was used to assess oral health-related quality of life, using a Likert format rated on a 5-point scale (0 not at all, 4 very much) for 14 questions, higher scores represent the poorer oral condition-related quality of life, with a minimum 0 points and maximum 56 points.

SECONDARY OUTCOMES:
Swallowing function assessment | The 1, 30, 90, and 120 days after recruitment. The investigators wanted to see if exercise would help oral muscle performance, there's a lack of data on this, so the investigator couldn't determine a change over time.
  This was assessed using a questionnaire with EAT-10 and DRACE indicators that can detect the initial risks of dysphagia. A Chinese version of Eat-10, a self-reported outcome instrument on swallowing function, consisted of 10 questions on a 5-point Likert scale, with a minimum of 0 points and a maximum of 40 points. Physical symptoms of chewing and swallowing disorders were assessed via the Dysphagia Risk Assessment of the Community-dwelling elderly persons (DRACE) questionnaire. DRACE, which was translated by the research team, included 12 variables involving chewing, swallowing, coughing problems, etc., based on a 3-level scale from 0 (never occurs) to 2 (occurs frequently), with a minimum of 0 points and a maximum of 24 points. For both questionnaires, higher scores represent poorer swallowing function.
DDK rate | The 1, 30, 90, and 120 days after recruitment. The investigators wanted to see if exercise would help oral muscle performance, there's a lack of data on this, so the investigator couldn't determine a change over time.
  Oral diadochokinesis (DDK) performance developed by HKU specifically in Cantonese or English (depends on participants' mother tongue) will be used. Participants will be instructed to repeat /pa/, /ta/, /ka/ as accurately and as quickly as the participants could within 10s respectively, and /pataka/ within 15s, at their normal speaking loudness level, speech recordings will be analyzed by speech therapist for speech motor assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Kit Hon Tsoi, PhD, Principal Investigator — Faculty of Dentistry, The University of Hong Kong
Locations (1):
- Faculty of Dentisry, the University of Hong Kong, Hong Kong, Hong Kong SAR, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data, study protocol, statistical analysis methods, and informed consent form can be requested after research is published from the principal investigator (jkhtsoi@hku.hk) who will coordinate with the study senior centers and hospital to ensure that any data sharing complies with the General Data Protection Regulations, the Hong Kong Personal Data (Privacy) Ordinance, and other legal agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: the data will be available after the results are released and published.
Access Criteria: requested from the principal investigator via email: jkhtsoi@hku.hk

REFERENCES:
- [Background] Johnston, L. What fast-ageing countries such as china tell us about our economic future. CommonWealth Magazine 2019.
- [Background] Libicki, M.C.; Shatz, H.J.; Taylor, J.E. The economic burden of aging populations. In Global demographic change and its implications for military power, RAND Corporation: 2011; pp 59-82.
- [Background] Hong kong population projections 2020-2069. The Government of HKSAR: Hong Kong, 2020.
- [Background] Rodrigues HL Jr, Scelza MF, Boaventura GT, Custodio SM, Moreira EA, Oliveira Dde L. Relation between oral health and nutritional condition in the elderly. J Appl Oral Sci. 2012 Feb;20(1):38-44. doi: 10.1590/s1678-77572012000100008. PMID 22437676
- [Background] Nitschke I, Muller F. The impact of oral health on the quality of life in the elderly. Oral Health Prev Dent. 2004;2 Suppl 1:271-5. PMID 15646585
- [Background] Pillai RS, Iyer K, Spin-Neto R, Kothari SF, Nielsen JF, Kothari M. Oral Health and Brain Injury: Causal or Casual Relation? Cerebrovasc Dis Extra. 2018;8(1):1-15. doi: 10.1159/000484989. Epub 2018 Jan 9. PMID 29402871
- [Background] Dominy SS, Lynch C, Ermini F, Benedyk M, Marczyk A, Konradi A, Nguyen M, Haditsch U, Raha D, Griffin C, Holsinger LJ, Arastu-Kapur S, Kaba S, Lee A, Ryder MI, Potempa B, Mydel P, Hellvard A, Adamowicz K, Hasturk H, Walker GD, Reynolds EC, Faull RLM, Curtis MA, Dragunow M, Potempa J. Porphyromonas gingivalis in Alzheimer's disease brains: Evidence for disease causation and treatment with small-molecule inhibitors. Sci Adv. 2019 Jan 23;5(1):eaau3333. doi: 10.1126/sciadv.aau3333. eCollection 2019 Jan. PMID 30746447
- [Background] Taghizadeh-Hesary, F.; Yoshino, N.; Mortha, A.; Taghizadeh-Hesary, F.; Roshanmehr, F.; Fiallos, J.; Tajra, E.; Bolanos, J.; Amaya, M.; Dang, J., et al. Economic burden of neurological disorders in an aging society (japan): A panel data analysis. . In ADBI Working Paper 1092, Asian Development Bank Institute: Tokyo, 2020.
- [Background] Yon, M.J.Y.; Lam, Y.H.W.; Tsoi, K.H. Do economic and dental resources affect older persons' ohrqol? In IADR/PER 96th General Session & Exhibition, International Association for Dental Research. The Abstract's web site is located at http://www.iadr.org/: United States, 2018; Vol. 97, p no. 3003.
- [Background] Miura, H.; Tano, T. Recent measures in geriatric oral health care in japan. J. Natl. Inst. Public Health 2019, 68, 8-16.
- [Result] O'Connor, S. (2014). World will have 13 'super-aged'nations by 2020. Financial Times, 11.